CLINICAL TRIAL: NCT03258385
Title: Effects of Vitamin B12 Fortified Milk Supplementation During Pregnancy and 6 Month Postpartum to Improve B12 Status and Child Development
Brief Title: Vitamin B12 Supplementation to Improve B12 Status and Child Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of California, Davis (Other); Nestlé Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: PR-16003
Record Dates: First submitted 2017-08-13; First posted 2017-08-23 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2021-04

CONDITIONS: Early Pregnancy
Keywords: Vitamin B12, Fortified milk, Immunity, Child development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin B12-fortified UHT milk (Active Comparator): Supplementation group (N=74) that will receive vitamin B12 fortified UHT milk daily
  Interventions: Dietary Supplement: Vitamin B12 fortified UHT milk
- Plain UHT milk (Placebo Comparator): Placebo group (N=74) that will receive plain UHT milk daily
  Interventions: Dietary Supplement: Plain UHT milk

INTERVENTIONS:
Dietary Supplement: Vitamin B12 fortified UHT milk — Daily intake of 200 mL of UHT milk fortified with 100 µg vitamin B12
  Arms: Vitamin B12-fortified UHT milk
Dietary Supplement: Plain UHT milk — Daily intake of 200 mL of plain UHT milk
  Arms: Plain UHT milk

SUMMARY:
Impaired vitamin B12 (B12) status during pregnancy is associated with increased risk of birth defects and common complications (e.g. intrauterine growth restriction, neural tube defects), and possibly immune function impairment. The newborns and infants of B12-deficient mothers have low B12 stores at birth, further exacerbated by a very low concentration of B12 in breast milk that may hinder their growth and development. In regions such as Bangladesh, many women of reproductive age have inadequate B12 status, probably due to low intake of animal source food. Vitamin B12 intake and status in pregnancy and lactation is potentially insufficient to prevent impaired child development and immune function related to inadequate B12 status. The investigators hypothesize that prolonged vitamin B12 supplementation through fortified milk starting from early pregnancy up to 6 mo-postpartum will improve: (1) biomarkers of vitamin B12 status in mothers-infant pairs (2) vaccine specific adaptive immunity in infants; (3) neurological and cognitive function in infants.

DETAILED DESCRIPTION:
The investigators aim to conduct a double-blind, randomized trial, to investigate the effects of B12-fortified milk on maternal and infant B12 status, immune function and child development. Pregnant women (n=148) will be randomized to receive B12-fortified milk (100 μg/day) or milk without fortification. The daily supplementation beginning at the baseline visit (GW 11-14) will continue until 6 mo-postpartum. Biomarkers of B12 status will be measured in mothers (GW 11-14 and 6-mo postpartum) and infants (3 and 6-mo). Infant development (6 and 12-mo) will be evaluated by Bayley Scales of Infant and Toddler Development. Immune responses will be measured in infant at 3 and 6-mo. Data on socioeconomic status, dietary diversity, and anthropometric indices will be recorded at baseline. Additional tests in mothers include screening for H. pylori and plasma gastrin.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 35 y old 2. 11-14 wk pregnant (based on last menstrual period) 3. Willing to stay in Dhaka during pregnancy and remain in the area for the 12 mo following recruitment 4. Willing to be admitted in the clinic for delivery 5. Intends to exclusively or predominantly breastfeed infant until 6 mo of age

-

Exclusion Criteria:

1. Women with severe anemia; Hb concentration <70 g/L 2. History or presence of systemic disease such as Diabetes mellitus, Hypertension 3. History of previous complicated pregnancies, pre-term delivery, or abortion 4. Current use of supplements containing vitamin B12 5. Children with acute illness or features suggestive of any chronic disease such as tuberculosis, any congenital anomalies such as cleft lip or palate.

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change in concentrations of biomarkers of vitamin B12 in mother-child pairs | Baseline and 6 months postpartum
  The investigators will determine the change in concentrations of biomarkers of B12 ( based on measurement of B12, MMA, tHcy, holoTC, cB12, folate in plasma; B12 in breast milk)
Vaccine specific immunity in infants | 6 months
  The investigators will determine the concentrations of vaccine specific IgA and IgG in plasma
Cognitive, Language and Motor Composite Score | 12 months
  The outcomes are measured by Bayley-III test
Nuroinflammatory cytokines | 12 months
  The investigators will determine the change in concentrations of EGF and TNF-α in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Towfida J Siddiqua, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Maternal and Child Health Training Institute, Dhaka, Bangladesh

REFERENCES:
- [Derived] Finkelstein JL, Fothergill A, Venkatramanan S, Layden AJ, Williams JL, Crider KS, Qi YP. Vitamin B12 supplementation during pregnancy for maternal and child health outcomes. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD013823. doi: 10.1002/14651858.CD013823.pub2. PMID 38189492